CLINICAL TRIAL: NCT06373744
Title: Metronomic Chemotherapy in a Real-world Population of Advanced Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Dr, Sun Yat-sen University
Other Study IDs: SYSU-022
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; metronomic chemotherapy; capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metronomic chemotherapy: Patients with advanced breast cancer who received metronomic chemotherapy.
  Interventions: Drug: cyclophosphamide , methotrexate , vinorelbine ,capecitabine

INTERVENTIONS:
Drug: cyclophosphamide , methotrexate , vinorelbine ,capecitabine — The drugs used in metronomic chemotherapy are cyclophosphamide (CTX), methotrexate (M), vinorelbine (VNR), and capecitabine

SUMMARY:
The goal of this observational study is to learn about the effects of metronomic chemotherapy in advanced breast cancer patients. The main question it aims to answer is:

How effective is metronomic chemotherapy in advanced breast cancer? Specific benefit groups of metronomic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Females, >18 years old;
2. Diagnosed with advanced breast cancer when using metronomic chemotherapy;
3. At least one clinical evaluation, including physical examination and imaging, according to the instructions of the supervising physician during the use of metronomic chemotherapy. Examinations include ultrasound, computed tomography, and magnetic resonance imaging;
4. Metronomic chemotherapy can be used alone, and patients who use it in combination with other drugs can also be included;
5. The clinical pathological information that needs to be collected is complete.

Exclusion Criteria:

1. Taking the drug for less than 2 weeks;
2. losing follow-up after taking the therapy;
3. The patient's breast cancer was still in the early stage when taking the therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced breast cancer taking metronomic chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to approximately 20 months
  Time from randomization to the first documentation of objective tumor progression or to death due to any cause without documented progression

SECONDARY OUTCOMES:
Overall Survival | Baseline until death (up to approximately 40 months)
  Time from randomization to date of death due to any cause
Objective Response Rate | Baseline up to approximately 20 months
  Objective response is defined as a complete response (CR) or partial response (PR) according to RECIST v.1.1. recorded from randomization until disease progression or death due to any cause.
Disease Control Rate | Baseline up to approximately 20 months
  Disease control is defined as complete response (CR), partial response (PR), or stable disease (SD) >24 weeks according to the RECIST version 1.1 recorded in the time period between randomization and disease progression or death to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Shusen Wang, Guangzhou, Gangdong, China

IPD SHARING:
Plan to Share IPD: Undecided